CLINICAL TRIAL: NCT04905095
Title: CSAPG Early Warning Score
Acronym: CEWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSAPG-11
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-03

CONDITIONS: Undefined
Keywords: Hospital Stay; Mortality; Clinical Deterioration
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EWS (Experimental): Early Warning Score will be implemented in the computer system of the nursing station
  Interventions: Other: EWS
- Control (Active Comparator): Nursing supervision will be carried out in the usual way.
  Interventions: Other: usual clinical care

INTERVENTIONS:
Other: EWS — Early Warning Score will be implemented in the computer system of the nursing station which belong to this intervention group. When the nurses enter the vital signs of the patients into the system, the EWS will be automatically calculated and an alarm will be displayed if an intervention is necessary, which is protocolized.
  Arms: EWS
Other: usual clinical care — Nurses perform their clinical monitoring activities as usual. EWS will not be implemented in their nursing station
  Arms: Control

SUMMARY:
The Early Warning Score (EWS) has been shown in previous studies to be correlated with mortality and mean hospital stay, but it is unknown whether the implementation of the scale improves mortality and mean hospital stay.

This trial aims to study whether the implantation of the EWS in a regional hospital reduces the mean hospital stay (primary objective), mortality and complications (secondary objectives).

For this, an open clinical trial will be carried out in which the hospitalization floors of the hospital will be administratively divided into two sections (two study branches); the EWS scale will be implemented in the computer equipment of one of the sections of each floor, acting the another section as a control branch.

All the patients admitted to the participating hospital floors during one year will be included in the study. The mean stay, mortality and complications will be compared between study branches.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted during study period to the participant hospital units.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15998 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital stay | from baseline to hospital discharge, as much 3 months
  Average days of hospital admission

SECONDARY OUTCOMES:
Mortality | from baseline to hospital discharge, as much 3 months
  Percentage of patients deceased during hospital admission
Complications | from baseline to hospital discharge, as much 3 months
  Percentage of patients who develop health complications during hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramos, Nurse, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari de l'Alt Penedès i Garraf, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.